CLINICAL TRIAL: NCT02267629
Title: Open Label Trial of Rapastinel (Formerly GLYX-13) in Individuals With Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6986
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — GLYX-13 peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental:Rapastinel (formerly GLYX-13) (Experimental): 10 mg/kg IV Rapastinel (formerly GLYX-13) infusion followed by assessments daily for a week, and weekly for a week.
  Interventions: Drug: Rapastinel (formerly GLYX-13)

INTERVENTIONS:
Drug: Rapastinel (formerly GLYX-13) — 10 mg/kg IV Rapastinel (formerly GLYX-13)

SUMMARY:
This research study tests whether GLYX-13 - an experimental drug that acts on a brain receptor called NMDA - can decrease symptoms of OCD within hours. This is not a treatment study. Results from this study will allow doctors and researchers to better understand if you and others with OCD may respond to a class of medications that target the NMDA brain receptor.

ELIGIBILITY:
Inclusion Criteria for Patients with No medication Washout:

* Age 18-55
* Physically healthy and not currently pregnant
* Primary Diagnosis of OCD
* currently off all psychotropic medications and other drugs
* Able to provide informed consent

Exclusion Criteria for Patients with No Medication Washout:

* Psychiatric conditions that make participation unsafe (schizophrenia [either self or first degree relative e.g. siblings, parents], history of violence, severe depression, eating disorder, substance abuse in prior year[including nicotine], lifetime substance dependence disorder [except nicotine])
* Female patients who are either pregnant or nursing
* Enrolled in or planning to enroll in Cognitive Behavioral Therapy.
* Medical conditions that make participation unsafe (e.g., high blood pressure, head injury)
* Currently on medications that make participation unsafe
* History of allergy, sensitivity, or intolerance to N-methyl-D-aspartate receptor (NMDAR) ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.

Inclusion Criteria for Patients with Medication Washout:

* Age 18-55
* Physically healthy and not currently pregnant
* Primary Diagnosis of OCD
* Currently on adequate dose of medication for treatment of OCD, but have not achieved at least partial remission and able to handle a medication washout.
* Able to provide informed consent

Exclusion Criteria for Patients with Medication Washout:

* Psychiatric conditions that make participation unsafe (schizophrenia [either self or first degree relative e.g. siblings, parents], history of violence, severe depression, eating disorder, substance abuse in prior year[including nicotine], lifetime substance dependence disorder [except nicotine])
* Female patients who are either pregnant or nursing
* Enrolled in or planning to enroll in Cognitive-Behavioral Therapy.
* Patient judged unlikely to be able to tolerated a medication washout.
* Medical conditions that make participation unsafe (e.g., high blood pressure, head injury)
* Currently on medications that make participation unsafe
* History of allergy, sensitivity, or intolerance to N-methyl-D-aspartate receptor (NMDAR) ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- New York State Psychiatric Insitute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez CI, Zwerling J, Kalanthroff E, Shen H, Filippou M, Jo B, Simpson HB, Burch RM, Moskal JR. Effect of a Novel NMDA Receptor Modulator, Rapastinel (Formerly GLYX-13), in OCD: Proof of Concept. Am J Psychiatry. 2016 Dec 1;173(12):1239-1241. doi: 10.1176/appi.ajp.2016.16080868. No abstract available. PMID 27903098
- See also: Website for Study — http://www.columbia-ocd.org
- See also: Rodriguez Lab - Stanford University — http://rodriguezlab.stanford.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental:Rapastinel (Formerly GLYX-13)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental:Rapastinel (Formerly GLYX-13)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Scores Change in Yale-Brown Obsessive Compulsive Challenge Scale (YBOCCS) Scores From Baseline to 230 Minutes Postinfusion.
Description: Patients self-rated the severity of their obsessions and compulsions using the YBOC Challenge Scale, a 10-item self-report form that assesses Obsessive Compulsive Disorder (OCD) symptoms (i.e., time spent, degree of control, severity) [total score range = 0 - 40 ] over the previous 60 minutes. The higher the number on the YBOCCS, the more severe the symptoms.
Time Frame: Baseline and 230 minutes post infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental:Rapastinel (Formerly GLYX-13)
Number analyzed (Participants) | 7
units on a scale | 13.71 (6.47)

2. Secondary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Yale-Brown Obsessive-Compulsive Scale.
Description: Patients given YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response was defined as at least a 35% reduction on the YBOCS.
Time Frame: Baseline and 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental:Rapastinel (Formerly GLYX-13)
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: over one week post infusion
Arm/Group | Experimental:Rapastinel (Formerly GLYX-13)
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No